CLINICAL TRIAL: NCT01567670
Title: Clinical Controlled Trial on Extinction of Opioidergic Binge Eating Disorder (BED) With Intranasal Naloxone Administration
Brief Title: Clinical Trial on Binge Eating Disorder, Treatment With Naloxone Spray
Acronym: BED
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lightlake Sinclair Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 72925
Record Dates: First submitted 2012-03-13; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naloxone (Active Comparator): nasal spray before binging, naloxone dose 2 mg, maximum daily dose 4 mg
  Interventions: Drug: Naloxone
- nasal spray (Placebo Comparator): nasal placebo (h2o) spray before binging, max sprays / day
  Interventions: Drug: naloxone placebo

INTERVENTIONS:
Drug: Naloxone — 2 mg x 1-2
  Arms: Naloxone
Drug: naloxone placebo — h2o placebo spray
  Arms: nasal spray

SUMMARY:
The investigators are studying a new treatment for one subtype of obesity. Obesity is not a disease. It is a symptom of several different diseases. These diseases have distinct etiologies, being caused by aberrations in different mechanisms. Forms of obesity caused by such non-critical mechanisms might be corrected fairly easily and safely. The investigators are interested in overeating and obesity that is caused by the opioidergic system. The opioidergic system appears to be responsible for a subtype of obesity associated with binge eating disorder (BED). People, especially with the right genetic predisposition, can become addicted to foods that release endorphins, in the way that people become addicted to exogenous opiates and other drugs that release endorphins. The particular application in our proposed clinical trial is for intranasal (IN) naloxone. The peak levels of naloxone were similar and the bioavailability of naloxone intranasally was 100% (the same) of that available IV." IN administration of naloxone has since been broadly tested in humans, as well, where it has been shown to be safe, with pharmacokinetics similar to those of naloxone given by injection .

ELIGIBILITY:
Inclusion Criteria:

* Binge eating disorder (DSM-IV) and body mass index (BMI) > 25
* Binge eating screen > 20

Exclusion Criteria:

* Pregnancy
* Drug usage
* Retarded
* Severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in frequency of binge eating | 0 and 24 week

SECONDARY OUTCOMES:
Becks depression inventory (BDI) | -1,0, 24 weeks
Analogic binge eating craving scale (BES-VAS) | -1,0,24 weeks
Binge eating severity scale (BES) | -1,0,24 weeks